CLINICAL TRIAL: NCT05883241
Title: Sustained Acoustic Medicine (SAM) for Symptomatic Treatment of Pain Related to Bone Fracture
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BF-01-2023
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Bone Fracture; Fresh Fracture
Keywords: Low-Intensity Ultrasound; Drug Delivery; Sonophoresis; Transdermal Drug Delivery; Non-Steroidal Anti-Inflammatory Drugs; Sustained Acoustic Medication; Low-Intensity Continuous Ultrasound
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SAM Ultrasound Device and Diclofenac Patch (Experimental): Patients receive treatment from the wired SAM Ultrasonic Diathermy Device for 4 hours at least 5 days a week for 12 weeks combined with 2.5% diclofenac patch. The SAM Device emits continuous ultrasound at 3-megahertz (MHz) frequency and 0.132 watts/cm^2 intensity.
  Interventions: Device: Sustained Acoustic Device with 2.5% Diclofenac Patch; Drug: 2.5% Diclofenac Patches

INTERVENTIONS:
Device: Sustained Acoustic Device with 2.5% Diclofenac Patch — Patients apply the SAM Ultrasonic Diathermy Device daily for 1-4 hours of continuous therapeutic ultrasound at 3-megahertz (MHz) frequency and 0.132 Watts/cm^2 with 2.5% Diclofenac patches.
  Other Names: ZetrOZ Ultrasound Device; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device Wearable; Long Duration Low-Intensity Device
Drug: 2.5% Diclofenac Patches — Topical pain relief-gel worn during treatment via SAM patch.

SUMMARY:
The purpose of this study is to assess the ability of long-duration low-intensity therapeutic ultrasound (LITUS) to alleviate bone-fracture related pain over a 12-week period.

The primary objective of this study is to evaluate the analgesic effect of LITUS in subjects suffering from bone-fracture pain.

Secondary objectives are to assess the ability of LITUS to improve patients return to work time.

DETAILED DESCRIPTION:
This is a 12-week study to clinically evaluate the effectiveness of the Sustained Acoustic Medicine (SAM) device combined with diclofenac on symptoms of patients suffering from pain related to a bone fracture(s). The class-II device, sam®, has been FDA-cleared for home use. On the first day of the study, baseline data will be collected as patients report pain score before treatment. During the following 12 weeks, patients will self-apply their treatment for the 4 hours daily. Each day of the study, pain scores will be recorded immediately before application of SAM device, during treatment, and at the completion of treatment.

Over 90 subjects will be recruited from neighboring communities to the study site(s). The study is designed to reach a diverse target patient population.

ELIGIBILITY:
Inclusion Criteria:

* Have physician-diagnosed bone fracture
* Are between 18-80 years of age
* Report a pain score between 3-7 (range: 0-10) prior to enrolment
* Report that pain from fracture negatively affects quality of life
* Are willing not to use any cream, gel, or topical solution during the administration of treatment other than the approved treatment provided to the subject at the initiation of the study
* Are deemed appropriate by their physician or by the study site physician to participate.
* Be willing and able to self-administer treatment daily within their place of residence or during normal daily activity, excluding bathing, showering, or other water activities which may result in submersion of the study device.
* Not use or initiate opioid and/or non-opioid analgesic medications.
* Be willing to discontinue any other interventional treatment modalities on the affected area during the study period (e.g., transcutaneous electrical nerve stimulation, electronic muscle stimulation, traditional ultrasound).

Exclusion Criteria:

* Cannot successfully demonstrate the ability to put on and take off the device.
* Displays any condition which, in the judgment of the investigator, would make participation in the study unacceptable including, but not limited to, the subject's ability to understand and follow instructions.
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening.
* Is pregnant.
* Is a prisoner.
* Is non-ambulatory (unable to walk).
* Has a pacemaker.
* Has a malignancy in the treatment area.
* Has an active infection, open sores, or wounds in the treatment area.
* Has impaired sensation in the treatment area, such as caused by chemotherapy or anesthesia.
* Has a known neuropathy (disease of the brain or spinal nerves).
* Has a hereditary disposition (tendency) for excessive bleeding (hemorrhage).
* Are currently taking steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Units on a Scale (0-10) 0 Being Least, 10 Being Worst Pain from Baseline | Through study completion, average of 12 weeks.
  Change in the self-described pain units on a scale by patient at baseline and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: George K. Lewis, Ph.D., Principal Investigator — ZetrOZ Systems
Locations (2):
- United States (2):
  - ZetrOZ Systems LLC, Trumbull, Connecticut
  - National Sports Medicine Institute, Lansdowne, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Class II Medical Device — https://samrecover.com